CLINICAL TRIAL: NCT02987023
Title: Uterus Transplantation From Live Donors With Robotic Assisted Surgery - Gothenburg II
Acronym: UTX-robot
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Brännström, Professor, Sahlgrenska University Hospital
Other Study IDs: SahlgrenskaUTx
Record Dates: First submitted 2016-11-29; First posted 2016-12-08 (Estimated); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Infertility, Female
Keywords: infertility, uterus, transplantation
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — blood, endometrial tissue, cervical tissue, placental tissue
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: uterus transplantation — Uterus transplantation from live donor

SUMMARY:
The study is a follow up of NCT01844362. Uterus transplantation will be performed from live donors to patients with uterine factor infertility. If will be performed before transplantation. Organ procurement from the donor will be performed by robotic assisted laparoscopy. Transplantation will be by laparotomy. Embryo transfer will be done 10-12 months after transplantation. After birth of 1-3 children the uterus will be removed by hysterectomy,

DETAILED DESCRIPTION:
The study is a follow up of NCT01844362. Uterus transplantation will be performed from live donors to patients with uterine factor infertility. If will be performed before transplantation. Organ procurement from the donor will be performed by robotic assisted laparoscopy. Transplantation will be by laparotomy. Embryo transfer will be done 10-12 months after transplantation. After birth of 1-3 children the uterus will be removed by hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* age below 38 years
* absolute uterine factor infertility
* BMI<30

Exclusion Criteria:

* systemic disease
* psychiatric disease

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: absolute uterine factor infertile women > 38 years
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-11; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Live births after uterus transplantation | 5 years
  Assessed by records from birthing unit and Swedish National Birth registry

SECONDARY OUTCOMES:
Development of children after uterus transplantation | 8 years
  Assessed by growth parameters and neuropsychiatric tests (Bayley Mental Scale, M-CHAT, CBCL, WPPSI-IV)

CONTACTS AND LOCATIONS:
Overall Officials: Mats Brännström, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared.

REFERENCES:
- [Background] Dahm-Kahler P, Kvarnstrom N, Brannstrom M. Robotic live donor hysterectomy. Curr Opin Organ Transplant. 2021 Dec 1;26(6):640-645. doi: 10.1097/MOT.0000000000000926. PMID 34593704
- [Background] Brannstrom M, Kvarnstrom N, Groth K, Akouri R, Wiman L, Enskog A, Dahm-Kahler P. Evolution of surgical steps in robotics-assisted donor surgery for uterus transplantation: results of the eight cases in the Swedish trial. Fertil Steril. 2020 Nov;114(5):1097-1107. doi: 10.1016/j.fertnstert.2020.05.027. Epub 2020 Aug 19. PMID 32828495
- [Background] Brannstrom M, Dahm-Kahler P, Ekberg J, Akouri R, Groth K, Enskog A, Broecker V, Molne J, Ayoubi JM, Kvarnstrom N. Outcome of Recipient Surgery and 6-Month Follow-Up of the Swedish Live Donor Robotic Uterus Transplantation Trial. J Clin Med. 2020 Jul 22;9(8):2338. doi: 10.3390/jcm9082338. PMID 32707899
- [Derived] Wentz E, Hagberg B, Hagberg H, Bokstrom H, Brannstrom M. Uterus transplantation; first data on neurologic, neuropsychiatric, and physical examination follow-up of children up to 6 years of age. Hum Reprod. 2025 Dec 1;40(12):2419-2429. doi: 10.1093/humrep/deaf178. PMID 40971624
- [Derived] Brannstrom M, Dahm-Kahler P, Kvarnstrom N, Enskog A, Olofsson JI, Olausson M, Molne J, Akouri R, Jarvholm S, Nilsson L, Stigson L, Hagberg H, Bokstrom H. Reproductive, obstetric, and long-term health outcome after uterus transplantation: results of the first clinical trial. Fertil Steril. 2022 Sep;118(3):576-585. doi: 10.1016/j.fertnstert.2022.05.017. Epub 2022 Jun 11. PMID 35697530